CLINICAL TRIAL: NCT02345733
Title: Use of a Novel Diet (UC DIET) Targeting the Microbiota for Treatment of Mild to Moderate Active Pediatric Ulcerative Colitis: An Open Label Pilot Study
Brief Title: Use of a Novel Diet (UC DIET) for Treatment of Mild to Moderate Active Pediatric Ulcerative Colitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prof. Arie Levine (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Arie Levine, Director, Pediatric Gastroenterology and Nutrition unit., Wolfson Medical Center
Organization: Wolfson Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0009-15-WOMC
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Doxycycline; Amoxicillin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ulcerative Colitis Diet (Experimental): Patients will receive a structured novel diet termed the UCD for 6 weeks, and those in remission at week 6 will receive the step down diet for another 6 weeks.
  Interventions: Other: Ulcerative Colitis Diet
- Antibiotic Treatment (Experimental): This antibiotic treatment will be given as an open label for patients who refuse diet therapy or for patients who show no improvement by week 3 , deteriorate by week 6, or patients who are not in full remission by week 6 will receive a 14 day course of antibiotics as previously described by Kato and colleagues.
  Interventions: Drug: Antibiotic cocktail

INTERVENTIONS:
Other: Ulcerative Colitis Diet — we have postulated that a diet that we developed that reduces exposure to dietary ingredients that allow sulfide reducing bacteria to thrive, or that impair the mucous layer, coupled with dietary products that enhance butyrate production, could induce remission in UC without involving additional immune suppression.
  Arms: Ulcerative Colitis Diet
Drug: Antibiotic cocktail — We have postulating that antibiotic therapy can alter the microbiota clinically. Controlling the microbiota by antibiotics may allow for control of the disease without immune suppression
  Other Names: •Doxycyclin, amoxicillin and metronidazole
  Arms: Antibiotic Treatment

SUMMARY:
The goal of the study is to evaluate strategies that target the microbiota for the treatment of Ulcerative Colitis , This study will involve a novel diet that the investigators developed , based on the hypothesis that UC involves dysbiosis , underutilzation of certain metabolic pathways and use of pathways that increase risk of inflammation . The investigators have postulated that manipulation of colonic bacterial metabolism with this diet will induce remission in UC without involving additional immune suppression.

DETAILED DESCRIPTION:
Ulcerative colitis is a chronic inflammatory disease primarily involving the colon. It has long been considered to be due to a dysregulated immune response targeting the colon, and involves unknown environmental factors . Recent studies have highlighted several characteristics which may suggest that UC is associated with alterations of the microbiota, defective production of short chain fatty acids and an impaired mucous layer. However at present, no effective therapy targets the microbiota or its interaction with the colonic epithelium. UC in humans is characterized by increased mucosal sulfides and increased sulfate and sulfide reducing bacteria and activation of amino acid metabolism pathways which impair butyrate production, whereas certain dietary patterns in humans and rodent models may induce dysbiosis and favor sulphide reducing bacteria. Further support for targeting the microbiota includes several studies demonstrating that antibiotics might be helpful for severe refractory colitis. Development of treatment strategies that target the microbiota could reduce exposure to immune suppression, and add new therapeutic strategies that do not exist at present.

Though diet has a significant impact on the composition of the microbiota no dietary intervention to date has proven effective for induction of remission. The investigators hypothesized that ulcerative colitis is caused by a series of events involving dysbiosis with sulfate or sulfide reducing bacteria combined with defective production of short chain fatty acids, coupled with a defective mucous layer.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Established diagnosis of UC.
3. Age: 8 - 19 years ( inclusive)
4. Mild to moderate active disease, 10 ≤ PUCAI ≤45.
5. Stable medication (IMM/ 5ASA) use for the past 6 weeks. Patients who have received topical 5ASA therapy for <7 days and are active may be included if topical therapy is stopped at enrolment

Exclusion Criteria:

Exclusion criteria:

1. Any proven current infection such as positive stool culture, parasite or C. difficile.
2. Antibiotic or Steroids use in the past 2 weeks.
3. PUCAI >45
4. Acute severe UC in the previous 12 months.
5. Current Extra intestinal manifestation of UC.
6. PSC or Liver disease
7. Pregnancy.
8. Allergy to one of the antibiotics or age <11 will exclude patients from entering the antibiotic arm

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Remission rate, defined as a PUCAI less than 10 at week 6. | week 6

SECONDARY OUTCOMES:
Mean PUCAI week 6 | week 6
Mean Calprotectin at week 6 | week 6
Physicians Global Assessment week 6 | week 6
Remission week 12, defined as a PUCAI less than 10 | week 12
Mean PUCAI week 12 | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Arie Levine, MD, Principal Investigator — Wolfson Medical Center
Locations (3):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States
- IWK Health Centre, Dalhousie University, Halifax, Nova Scotia, Canada
- The E. Wolfson.Medical Center, Holon, Israel